CLINICAL TRIAL: NCT04885530
Title: ACTIV-6: COVID-19 Outpatient Randomized Trial to Evaluate Efficacy of Repurposed Medications
Brief Title: ACTIV-6: COVID-19 Study of Repurposed Medications
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Susanna Naggie, MD (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Susanna Naggie, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00107921; 3U24TR001608-05W1 (NIH)
Record Dates: First submitted 2021-04-30; First posted 2021-05-13 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Covid19
Keywords: SARS-CoV-2; COVID-19; ivermectin; Placebo; Duke University Health System; Outcomes; Duke Clinical Research Institute; fluticasone; fluvoxamine; ACTIV 6; ACTIV; montelukast; metformin
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Fluvoxamine; Fluticasone; fluticasone furoate; montelukast; Metformin

STUDY DESIGN:
Intervention Model Description: Double-Blind, Placebo-Controlled, Randomized Trial
Who Masked: Participant, Care Provider
Masking Description: The participant and study teams will know which study drug the participant is allocated to, but will be blinded to study drug versus placebo because they will be matching.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Arm A - Ivermectin 400 (Experimental): Ivermectin - 7-mg tablets
  Participant will be instructed to take a pre-specified number of tablets for 3 consecutive days based on their weight for a daily dose of approximately 300-400 µg/kg.
  Interventions: Drug: Ivermectin
- Arm A - Placebo (Placebo Comparator): Placebo - appearance and size matched to active study drug.
  Participant will be instructed to take a pre-specified number of tablets for 3 consecutive days based on their weight, matched to active study drug dosing.
  Interventions: Other: Placebo
- Arm B - Fluvoxamine (Experimental): Fluvoxamine will be self-administered orally by each participant at a dose of 50 mg twice a day for 10 days.
  Interventions: Drug: Fluvoxamine
- Arm B- Placebo (Placebo Comparator): Placebo - appearance and size matched to active study drug. Placebo will be self-administered orally by each participant twice a day for 10 days.
  Interventions: Other: Placebo
- Arm C - Fluticasone (Experimental): Fluticasone is a self-administered inhaled drug. Participants will self-administer 200 µg (1 blister) of fluticasone once daily for 14 days. After inhaler activation, the powder within the blister is exposed and the participant inhales the study drug through the mouthpiece.
  Interventions: Drug: Fluticasone
- Arm C - Placebo (Placebo Comparator): Placebo is a self-administered by inhalation. Participants will self-administer 1 blister of placebo once daily for 14 days. After inhaler activation, the powder within the blister is exposed and the participant inhales the placebo through the mouthpiece.
  Interventions: Other: Placebo
- Arm D - Ivermectin 600 (Experimental): Ivermectin - 7-mg tablets
  Participant will be instructed to take a pre-specified number of tablets for 6 consecutive days based on their weight for a daily dose of approximately 400-600 µg/kg.
  Interventions: Drug: Ivermectin
- Arm D - Placebo (Placebo Comparator): Placebo - appearance and size matched to active study drug.
  Participant will be instructed to take a pre-specified number of tablets for 6 consecutive days based on their weight, matched to active study drug dosing.
  Interventions: Other: Placebo
- Arm E - Fluvoxamine 100 (Experimental): Fluvoxamine will be self-administered orally by each participant at a dose of 50 mg twice a day for 1 day, followed by a dose of 100 mg twice a day for 12 days.
  Interventions: Drug: Fluvoxamine
- Arm E - Placebo (Placebo Comparator): Placebo - appearance and size matched to active study drug.
  Placebo will be self-administered orally by each participant, with number of tablets matched to active study drug dosing.
  Interventions: Other: Placebo
- Arm F - Montelukast (Experimental): Montelukast will be self-administered orally by each participant at a dose of 10 mg once a day for 14 days.
  Interventions: Drug: Montelukast
- Arm F - Placebo (Placebo Comparator): Placebo - appearance and size matched to active study drug.
  Placebo will be self-administered orally by each participant, with number of tablets matched to active study drug dosing.
  Interventions: Other: Placebo
- Arm G - Metformin (Experimental): Metformin IR tablets will be self-administered orally according to the following dosing schedule:
  * 500 mg on Day 1;
  * 500 mg in the morning and 500 mg in the evening on Day 2 through Day 5; and
  * 500 mg in the morning and 2 x 500 mg (a total of 1000 mg) in the evening on Day 6 through Day 14.
  Interventions: Drug: Metformin
- Arm G - Placebo (Placebo Comparator): Placebo - appearance and size matched to active study drug.
  Placebo will be self-administered orally by each participant, with number of tablets matched to active study drug dosing.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ivermectin — Each participant will receive a sufficient quantity of 7-mg tablets to be taken as directed based on their weight. The tablets are white, round, biconvex tablets with "123" over the scoring on one side. All packaging will be labeled to indicate that the product is for investigational use.
  Other Names: Ivermectin Tablets
  Arms: Arm A - Ivermectin 400; Arm D - Ivermectin 600
Drug: Fluvoxamine — Fluvoxamine is a round golden 50 mg tablet that is scored on both sides - one side has "APO" and the other side has "F50" with a partial bisect. All packaging will be labeled to indicate that the product is for investigational use, administered at a dose of 50 mg, twice daily for 10 days.
  Other Names: Fluvoxamine Maleate Tablets
  Arms: Arm B - Fluvoxamine; Arm E - Fluvoxamine 100
Drug: Fluticasone — Fluticasone furoate is an inhaled powder drug product composed of fluticasone furoate. It is a synthetic trifluorinated corticosteroid that is insoluble in water. Fluticasone furoate is a white powder and will be provided in a two tone grey inhaler with a mouthpiece cover and separate foil blister strips. The inhaler will be packaged in a moisture-protective foil tray with a desiccant and a peelable lid.All packaging will be labeled to indicate that the product is for investigational use. Participants will self-administer 200 µg (1 blister) of fluticasone furoate once daily for 14 days.
  Other Names: Fluticasone Furoate
  Arms: Arm C - Fluticasone
Other: Placebo — Each study arm will contain a placebo comparator. Placebo will look similar to study drug and will be administered via the same route of administration and dose. However, placebo will be an inactive substance, containing no study drug.
  Arms: Arm A - Placebo; Arm B- Placebo; Arm C - Placebo; Arm D - Placebo; Arm E - Placebo; Arm F - Placebo; Arm G - Placebo
Drug: Montelukast — Montelukast sodium is a white to off-white powder. The 10 mg montelukast tablets are beige, rounded square-shaped, biconvex, film-coated tablets. Each tablet contains 10.4 mg of montelukast sodium, which is equivalent to 10 mg montelukast. All packaging will be labeled to indicate that the product is for investigational use.
  Arms: Arm F - Montelukast
Drug: Metformin — Metformin IR tablets contain the active metformin hydrochloride and inactive ingredients including povidone and magnesium stearate. Commercially available metformin 500 mg tablets will be provided.
  Arms: Arm G - Metformin

SUMMARY:
The purpose of this study is to evaluate the effectiveness of repurposed medications (study drug(s) in reducing symptoms of non-hospitalized participants with mild to moderate COVID-19. Participants will receive either study drug or placebo. They will self-report any new or worsening symptoms or medical events they may experience while taking study drug or placebo. This study is intended to be all remote with no in person visits, unless the study team feels it is in the best interest of a participant to see them in person.

Prior and current drug arms are listed on clinicaltrials.gov and will be updated with the activation of any new drug arms. Each study arm will also have its own clinicaltrials.gov entry and will include "Pro00107921" in the Unique Protocol ID.

Pro00107921_A - Arm D (Ivermectin 400) - NCT05736861; Pro00107921_B - Arm B (Fluvoxamine) - NCT05890586; Pro00107921_C - Arm C (Fluticasone) - NCT05736874; Pro00107921_D - Arm D (Ivermectin 600) - NCT05894538; Pro00107921_E - Arm E (Fluvoxamine 100) - NCT05894564; Pro00107921_F - Arm F (Montelukast) - NCT05894577; Pro00107921_G - Arm G (Metformin) - NCT06042855.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a novel betacoronavirus that first emerged in December 2019 and has since caused a global pandemic unseen in almost a century with respect to the number of cases and overall mortality. The clinical disease related to SARS-CoV-2 is referred to as Coronavirus Disease 2019 (COVID-19). Over 2020, advances were made for treatment of COVID-19 and several vaccinations have received emergency use authorization for prevention of SARS-CoV-2 infections. However, the pandemic continues to evolve with new variants and surges of infections in different regions of the world, requiring an ongoing evidence-generating platform, in particular for the treatment of COVID-19 infection in the outpatient setting.

This proposed platform protocol can serve as an evidence generating system for prioritized drugs repurposed from other indications with an established safety record and preliminary evidence of clinical efficacy for the treatment of COVID-19. The ultimate goal is to evaluate if repurposed medications can make participants feel better faster and reduce death and hospitalization.

This platform protocol is designed to be flexible so that it is suitable for a wide range of settings within healthcare systems and in community settings where it can be integrated into routine COVID-19 testing programs and subsequent treatment plans. This platform protocol will enroll participants in an outpatient setting with a confirmed polymerase chain reaction (PCR) or antigen test for SARS-CoV-2.

Participants will be randomized to study drugs or placebo based on the arms that are actively enrolling at the time of randomization. Study drugs may be added or removed according to adaptive design and/or emerging evidence. When there are multiple study drugs available, randomization will occur based on appropriateness of each drug for the participant as determined by the study protocol and investigator and participant equipoise. Each participant will be required to randomize to at least one study drug versus placebo. The probability of placebo to treatment will remain the same regardless of eligibility decisions.

Eligible participants will be randomized (1:1), in a blinded fashion, to either the study drug arm or placebo arm in addition to standard of care. As additional study drugs are added, the randomization will be altered to leverage placebo data across arms. Participants will receive a complete supply study drug or placebo with the quantity depending on the study drug/placebo to which they are randomized.

All study visits are designed to be remote. However, screening and enrollment may occur in-person at sites and unplanned study visits may occur in-person or remotely, as deemed appropriate by the site investigator for safety purposes. Participants will be asked to complete questionnaires and report safety events during the study. Participants will be prompted by the online system to report safety events and these will be reviewed and confirmed via medical records and site staff, as necessary.

ELIGIBILITY:
Eligibility for overall study are listed below. There may be additional appendix-specific criteria.

Inclusion Criteria:

* Completed Informed Consent
* Age ≥ 30 years old
* Confirmed SARS-CoV-2 infection by any authorized or approved polymerase chain reaction (PCR) or antigen test collected within 10 days of screening
* Two or more current symptoms of acute infection for ≤7 days. Symptoms include the following: fatigue, dyspnea, fever, cough, nausea, vomiting, diarrhea, body aches, chills, headache, sore throat, nasal symptoms, new loss of sense of taste or smell

Exclusion Criteria:

* Current or recent (within 10 days of screening) hospitalization for COVID-19 infection
* Current or planned participation in another interventional trial to treat COVID-19, at the discretion of the study principal investigator (PI)
* Current or recent use (within the last 14 days) of study drug or study drug/device combination
* Known allergy/sensitivity or any hypersensitivity to components of the study drug or placebo
* Known contraindication(s) to study drug including prohibited concomitant medications
* Previous or current enrollment in the ACTIV-6 trial

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10956 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Naggie, MD, Principal Investigator — Duke Clinical Research Institute; Adrian Hernandez, MD, Principal Investigator — Duke Clinical Research Institute
Locations (110):
- United States (110):
  - Chandler Regional Medical Center, Chandler, Arizona
  - Lamb Health, LLC, Gilbert, Arizona
  - First Care Medical Clinic, Mesa, Arizona
  - Trident Health Center, Peoria, Arizona
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Assuta Family Medical Group APMC, North Hollywood, California
  - Stanford, Palo Alto, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Doctors Medical Group of Colorado Springs, P.C., Colorado Springs, Colorado
  - Pine Ridge Family Medicine Inc., Colorado Springs, Colorado
  - Tabitha B. Fortt, M.D., LLC, Stamford, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Arena Medical Group, Deerfield Beach, Florida
  - Lupus Foundation of Gainesville, Gainesville, Florida
  - University of Florida Health, Gainesville, Florida
  - L and A Morales Healthcare, Inc, Hialeah, Florida
  - University of Florida-JAX-ASCENT, Jacksonville, Florida
  - AMRON Vitality and Wellness Center, LLC, Jacksonville, Florida
  - Sunshine Walk In Clinic, Lake Mary, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Well Pharma Medical Research, Miami, Florida
  - The Angel Medical Research Corporation, Miami Lakes, Florida
  - Innovation Clinical Trials Inc., Palmetto Bay, Florida
  - Lice Source Services Plantation, Plantation, Florida
  - Premier Health, St. Petersburg, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - UF Health Precision Health Research, The Villages, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory Healthcare, Atlanta, Georgia
  - Essential Medical Care, Inc., College Park, Georgia
  - Clincept, LLC, Columbus, Georgia
  - HOPE Clinical Research and Wellness, Conyers, Georgia
  - David Kavtaradze MD, Inc., Cordele, Georgia
  - Elite Family Practice, Douglasville, Georgia
  - Christ the King Health Care, P.C., Loganville, Georgia
  - Miller Family Practice, LLC, Macon, Georgia
  - Northwestern Univesity, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Olivo Wellness Medical Center, Chicago, Illinois
  - NorthShore Medical Group, Evanston, Illinois
  - Advanced Medical Care, Ltd, Lake Zurich, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Franciscan Health Michigan City, Michigan City, Indiana
  - Del Pilar Medical and Urgent Care, Mishawaka, Indiana
  - University of Kansas - Wichita, Wichita, Kansas
  - A New Start II, LLC, Central City, Kentucky
  - Christus Saint Frances Hospita, Alexandria, Louisiana
  - University Medical Center- New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Jadestone Clinical Research, LLC, Rockville, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Health Quality Primary Care, Lawrence, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Ananda Medical Clinic, Dearborn, Michigan
  - GFC of Southeastern Michigan, PC, Detroit, Michigan
  - Romancare Health Services, Detroit, Michigan
  - Essentia Health, Duluth, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri - Columbia, Columbia, Missouri
  - Comprehensive Pain Management and Endocrinology, Henderson, Nevada
  - Focus Clinical Research Solutions, Bayonne, New Jersey
  - Raritan Bay Primary Care & Cardiology Associates, Matawan, New Jersey
  - G&S Medical Associates, LLC, Paterson, New Jersey
  - Mediversity Healthcare, Turnersville, New Jersey
  - Christus St. Vincent Regional Medical Center, Santa Fe, New Mexico
  - Geriatrics and Medical Associates, Clinton, New York
  - Weill Cornell Medical College, New York, New York
  - Spinal Pain and Medical Rehab, PC, Yonkers, New York
  - Vaidya MD PLLC, Clayton, North Carolina
  - Maria Medical Center, PLLC, Dunn, North Carolina
  - Duke Clinical Research Institute, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Lapis Clinical Research, Mooresville, North Carolina
  - Superior Clinical Research, Smithfield, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Diabetes and Endocrinology Assoc. of Stark County, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - TriHealth, Inc, Montgomery, Ohio
  - The Heart and Medical Center, Durant, Oklahoma
  - Hugo Medical clinic, Hugo, Oklahoma
  - Ascension St. John, Tulsa, Oklahoma
  - Bucks County Clinical Research, Morrisville, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinical Trials Center of Middle TN, Franklin, Tennessee
  - Rapha Family Wellness, Hendersonville, Tennessee
  - Medical Specialists of Knoxville, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Express Family Clinic, Allen, Texas
  - DHR Health Institute for Research, Edinburg, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Health Physicians Group, Fort Worth, Texas
  - Highlands Medical Associates, P.A., Highlands, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Family Practice Doctors P.A., Humble, Texas
  - Texas Health Physicians Group, Irving, Texas
  - Kintex Group Texas LLC, DBA Activian Clinical Research, Kingwood, Texas
  - University Diagnostics and Treatment Clinic, Pasadena, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Jeremy W. Szeto, D.O., P.A., Sugar Land, Texas
  - University of Texas Rio Grande Valley, Weslaco, Texas
  - University of Virginia, Charlottesville, Virginia
  - Providence Medical Research Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will share this data after it has been de-identified. We will share data beginning around 6 months after publication and for up to 36 months afterward. Access will only be shared with those who have obtained prior IRB approval to be able to access this data.
Supporting Information: SAP, CSR
Time Frame: Up to 36 months after publication
Access Criteria: Interested investigators will need to seek prior IRB approval before access to any data is granted.

REFERENCES:
- [Derived] Bramante CT, Stewart TG, Boulware DR, McCarthy MW, Gao Y, Rothman RL, Mourad A, Thicklin F, Cohen JB, Garcia Del Sol IT, Ruiz-Unger J, Shah NS, Mehta M, Cardona OQ, Scott J, Ginde AA, Castro M, Jayaweera D, Sulkowski M, Gentile N, McTigue K, Felker GM, Collins S, Dunsmore SE, Adam SJ, Lindsell CJ, Hernandez AF, Naggie S; Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group and Investigators. Metformin on Time to Sustained Recovery in Adults with COVID-19: The ACTIV-6 Randomized Clinical Trial. medRxiv [Preprint]. 2025 Jan 14:2025.01.13.25320485. doi: 10.1101/2025.01.13.25320485. PMID 41030935
- [Derived] Bramante CT, Stewart TG, Boulware DR, McCarthy MW, Gao Y, Rothman RL, Mourad A, Thicklin F, Cohen JB, Garcia Del Sol IT, Shah NS, Mehta M, Quintero Cardona O, Scott J, Ginde AA, Castro M, Jayaweera D, Sulkowski M, Gentile N, McTigue K, Felker GM, Collins S, Dunsmore SE, Adam SJ, Lindsell CJ, Hernandez AF, Naggie S; Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group and Investigators. Metformin on the Presence of COVID-19 Symptoms Over 6 Months: The ACTIV-6 Randomized Clinical Trial. medRxiv [Preprint]. 2025 Aug 12:2025.08.08.25333305. doi: 10.1101/2025.08.08.25333305. PMID 40832427
- [Derived] Bramante CT, Stewart TG, Boulware DR, McCarthy MW, Gao Y, Rothman RL, Mourad A, Thicklin F, Cohen JB, Garcia Del Sol IT, Ruiz-Unger J, Shah NS, Mehta M, Cardona OQ, Scott J, Ginde AA, Castro M, Jayaweera D, Sulkowski M, Gentile N, McTigue K, Felker GM, Collins S, Dunsmore SE, Adam SJ, Lindsell CJ, Hernandez AF, Naggie S; Accelerating COVID-19 Therapeutic Interventions and Vaccines-6 Study Group and Investigators. Metformin and Time to Sustained Recovery in Adults With COVID-19: The ACTIV-6 Randomized Clinical Trial. JAMA Intern Med. 2025 Sep 1;185(9):1092-1101. doi: 10.1001/jamainternmed.2025.2570. PMID 40658388
- [Derived] Rothman RL, Stewart TG, Mourad A, Boulware DR, McCarthy MW, Thicklin F, Garcia Del Sol IT, Garcia JL, Bramante CT, Shah NS, Singh U, Williamson JC, Rebolledo PA, Jagannathan P, Schwasinger-Schmidt T, Ginde AA, Castro M, Jayaweera D, Sulkowski M, Gentile N, McTigue K, Felker GM, DeLong A, Wilder R, Collins S, Dunsmore SE, Adam SJ, Hanna GJ, Shenkman E, Hernandez AF, Naggie S, Lindsell CJ; Accelerating COVID-19 Therapeutic Interventions and Vaccines-6 Study Group and Investigators. Time to Sustained Recovery Among Outpatients With COVID-19 Receiving Montelukast vs Placebo: The ACTIV-6 Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2439332. doi: 10.1001/jamanetworkopen.2024.39332. PMID 39422912
- [Derived] Rothman RL, Stewart TG, Mourad A, Boulware DR, McCarthy MW, Thicklin F, Garcia Del Sol IT, Garcia JL, Bramante CT, Shah NS, Singh U, Williamson JC, Rebolledo PA, Jagannathan P, Schwasinger-Schmidt T, Ginde AA, Castro M, Jayaweera D, Sulkowski M, Gentile N, McTigue K, Felker GM, DeLong A, Wilder R, Collins S, Dunsmore SE, Adam SJ, Hanna GJ, Shenkman E, Hernandez AF, Naggie S, Lindsell CJ; Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group and Investigators. Effect of Montelukast vs Placebo on Time to Sustained Recovery in Outpatients with COVID-19: The ACTIV-6 Randomized Clinical Trial. medRxiv [Preprint]. 2024 May 18:2024.05.16.24307115. doi: 10.1101/2024.05.16.24307115. PMID 38798524
- [Derived] Stewart TG, Rebolledo PA, Mourad A, Lindsell CJ, Boulware DR, McCarthy MW, Thicklin F, Garcia Del Sol IT, Bramante CT, Lenert LA, Lim S, Williamson JC, Cardona OQ, Scott J, Schwasinger-Schmidt T, Ginde AA, Castro M, Jayaweera D, Sulkowski M, Gentile N, McTigue K, Felker GM, DeLong A, Wilder R, Rothman RL, Collins S, Dunsmore SE, Adam SJ, Hanna GJ, Shenkman E, Hernandez AF, Naggie S; Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group and Investigators. Higher-Dose Fluvoxamine and Time to Sustained Recovery in Outpatients With COVID-19: The ACTIV-6 Randomized Clinical Trial. JAMA. 2023 Dec 26;330(24):2354-2363. doi: 10.1001/jama.2023.23363. PMID 37976072
- [Derived] Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group and Investigators; Naggie S. Effect of Higher-Dose Fluvoxamine vs Placebo on Time to Sustained Recovery in Outpatients with Mild to Moderate COVID-19: A Randomized Clinical Trial. medRxiv [Preprint]. 2023 Sep 13:2023.09.12.23295424. doi: 10.1101/2023.09.12.23295424. PMID 37745371
- [Derived] Boulware DR, Lindsell CJ, Stewart TG, Hernandez AF, Collins S, McCarthy MW, Jayaweera D, Gentile N, Castro M, Sulkowski M, McTigue K, Felker GM, Ginde AA, Dunsmore SE, Adam SJ, DeLong A, Hanna G, Remaly A, Thicklin F, Wilder R, Wilson S, Shenkman E, Naggie S; ACTIV-6 Study Group and Investigators. Inhaled Fluticasone Furoate for Outpatient Treatment of Covid-19. N Engl J Med. 2023 Sep 21;389(12):1085-1095. doi: 10.1056/NEJMoa2209421. PMID 37733308
- [Derived] Naggie S, Boulware DR, Lindsell CJ, Stewart TG, Slandzicki AJ, Lim SC, Cohen J, Kavtaradze D, Amon AP, Gabriel A, Gentile N, Felker GM, Jayaweera D, McCarthy MW, Sulkowski M, Rothman RL, Wilson S, DeLong A, Remaly A, Wilder R, Collins S, Dunsmore SE, Adam SJ, Thicklin F, Hanna GJ, Ginde AA, Castro M, McTigue K, Shenkman E, Hernandez AF; Accelerating Covid-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group and Investigators. Effect of Higher-Dose Ivermectin for 6 Days vs Placebo on Time to Sustained Recovery in Outpatients With COVID-19: A Randomized Clinical Trial. JAMA. 2023 Mar 21;329(11):888-897. doi: 10.1001/jama.2023.1650. PMID 36807465
- [Derived] McCarthy MW, Naggie S, Boulware DR, Lindsell CJ, Stewart TG, Felker GM, Jayaweera D, Sulkowski M, Gentile N, Bramante C, Singh U, Dolor RJ, Ruiz-Unger J, Wilson S, DeLong A, Remaly A, Wilder R, Collins S, Dunsmore SE, Adam SJ, Thicklin F, Hanna G, Ginde AA, Castro M, McTigue K, Shenkman E, Hernandez AF; Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group and Investigators. Effect of Fluvoxamine vs Placebo on Time to Sustained Recovery in Outpatients With Mild to Moderate COVID-19: A Randomized Clinical Trial. JAMA. 2023 Jan 24;329(4):296-305. doi: 10.1001/jama.2022.24100. PMID 36633838
- [Derived] Naggie S, Boulware DR, Lindsell CJ, Stewart TG, Lim SC, Cohen J, Kavtaradze D, Amon AP, Gabriel A, Gentile N, Felker GM, Rothman RL, Jayaweera D, McCarthy MW, Sulkowski M, Wilson S, DeLong A, Remaly A, Wilder R, Collins S, Dunsmore SE, Adam SJ, Thicklin F, Hanna GJ, Ginde AA, Castro M, McTigue K, Shenkman E, Hernandez AF; Accelerating Covid-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group and Investigators. Effect of Ivermectin 600 mug/kg for 6 days vs Placebo on Time to Sustained Recovery in Outpatients with Mild to Moderate COVID-19: A Randomized Clinical Trial. medRxiv [Preprint]. 2022 Dec 15:2022.12.15.22283488. doi: 10.1101/2022.12.15.22283488. PMID 36561174
- [Derived] Naggie S, Boulware DR, Lindsell CJ, Stewart TG, Gentile N, Collins S, McCarthy MW, Jayaweera D, Castro M, Sulkowski M, McTigue K, Thicklin F, Felker GM, Ginde AA, Bramante CT, Slandzicki AJ, Gabriel A, Shah NS, Lenert LA, Dunsmore SE, Adam SJ, DeLong A, Hanna G, Remaly A, Wilder R, Wilson S, Shenkman E, Hernandez AF; Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV-6) Study Group and Investigators. Effect of Ivermectin vs Placebo on Time to Sustained Recovery in Outpatients With Mild to Moderate COVID-19: A Randomized Clinical Trial. JAMA. 2022 Oct 25;328(16):1595-1603. doi: 10.1001/jama.2022.18590. PMID 36269852
- [Derived] Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group; Naggie S. Ivermectin for Treatment of Mild-to-Moderate COVID-19 in the Outpatient Setting: A Decentralized, Placebo-controlled, Randomized, Platform Clinical Trial. medRxiv [Preprint]. 2022 Aug 11:2022.06.10.22276252. doi: 10.1101/2022.06.10.22276252. PMID 35982669
- [Derived] Accelerating Covid-19 Therapeutic Interventions and Vaccines (ACTIV)-6 Study Group; Naggie S. Inhaled Fluticasone for Outpatient Treatment of Covid-19: A Decentralized, Placebo-controlled, Randomized, Platform Clinical Trial. medRxiv [Preprint]. 2022 Aug 11:2022.07.12.22277548. doi: 10.1101/2022.07.12.22277548. PMID 35982649
- [Derived] Dodds MG, Doyle EB, Reiersen AM, Brown F, Rayner CR. Fluvoxamine for the treatment of COVID-19. Lancet Glob Health. 2022 Mar;10(3):e332. doi: 10.1016/S2214-109X(22)00006-7. No abstract available. PMID 35180412

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Numbers reported represent those who were eligible for study drug and randomized. Participants who were randomized to a placebo group may have participated in more than one study arm due to the nature of the study design.
Groups:
- Arm A - Ivermectin 400: Ivermectin - 7-mg tablets or Placebo
  Participant will be instructed to take a pre-specified number of tablets for 3 consecutive days based on their weight for a daily dose of approximately 300-400 µg/kg.
  Ivermectin: Each participant will receive a sufficient quantity of 7-mg tablets to be taken as directed based on their weight. The tablets are white, round, biconvex tablets with "123" over the scoring on one side. All packaging will be labeled to indicate that the product is for investigational use.
- Arm B - Fluvoxamine: Fluvoxamine or Placebo will be self-administered orally by each participant at a dose of 50 mg twice a day for 10 days.
  Fluvoxamine: Fluvoxamine is a round golden 50 mg tablet that is scored on both sides - one side has "APO" and the other side has "F50" with a partial bisect. All packaging will be labeled to indicate that the product is for investigational use, administered at a dose of 50 mg, twice daily for 10 days.
- Arm C - Fluticasone: Fluticasone or Placebo is a self-administered inhaled drug. Participants will self-administer 200 µg (1 blister) of fluticasone once daily for 14 days. After inhaler activation, the powder within the blister is exposed and the participant inhales the study drug through the mouthpiece.
  Fluticasone: Fluticasone furoate is an inhaled powder drug product composed of fluticasone furoate. It is a synthetic trifluorinated corticosteroid that is insoluble in water. Fluticasone furoate is a white powder and will be provided in a two tone grey inhaler with a mouthpiece cover and separate foil blister strips. The inhaler will be packaged in a moisture-protective foil tray with a desiccant and a peelable lid.All packaging will be labeled to indicate that the product is for investigational use. Participants will self-administer 200 µg (1 blister) of fluticasone furoate once daily for 14 days.
- Arm D - Ivermectin 600: Ivermectin - 7-mg tablets or Placebo
  Participant will be instructed to take a pre-specified number of tablets for 6 consecutive days based on their weight for a daily dose of approximately 400-600 µg/kg.
  Ivermectin: Each participant will receive a sufficient quantity of 7-mg tablets to be taken as directed based on their weight. The tablets are white, round, biconvex tablets with "123" over the scoring on one side. All packaging will be labeled to indicate that the product is for investigational use.
- Arm E - Fluvoxamine 100: Fluvoxamine or Placebo will be self-administered orally by each participant at a dose of 50 mg twice a day for 1 day, followed by a dose of 100 mg twice a day for 12 days.
  Fluvoxamine: Fluvoxamine is a round golden 50 mg tablet that is scored on both sides - one side has "APO" and the other side has "F50" with a partial bisect. All packaging will be labeled to indicate that the product is for investigational use, administered at a dose of 50 mg, twice daily for 10 days.
- Arm F - Montelukast: Montelukast or Placebo will be self-administered orally by each participant at a dose of 10 mg once a day for 14 days.
  Montelukast: Montelukast sodium is a white to off-white powder. The 10 mg montelukast tablets are beige, rounded square-shaped, biconvex, film-coated tablets. Each tablet contains 10.4 mg of montelukast sodium, which is equivalent to 10 mg montelukast. All packaging will be labeled to indicate that the product is for investigational use.
- Arm G - Metformin: Metformin IR tablets or Placebo will be self-administered orally according to the following dosing schedule:
  * 500 mg on Day 1;
  * 500 mg in the morning and 500 mg in the evening on Day 2 through Day 5; and
  * 500 mg in the morning and 2 x 500 mg (a total of 1000 mg) in the evening on Day 6 through Day 14.
  Metformin: Metformin IR tablets contain the active metformin hydrochloride and inactive ingredients including povidone and magnesium stearate. Commercially available metformin 500 mg tablets will be provided.
Period: Substudy A
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin
Started | 1800 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1800 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy B
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin
Started | 0 | 1331 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 1331 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy C
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin
Started | 0 | 0 | 1407 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 1407 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy D
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin
Started | 0 | 0 | 0 | 1459 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 1459 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy E
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin
Started | 0 | 0 | 0 | 0 | 1208 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 1208 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy F
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin
Started | 0 | 0 | 0 | 0 | 0 | 1453 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 1453 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy G
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3214
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3214
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Numbers reported represent those who were eligible for study drug and randomized to each appendix.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin | Total
Number analyzed (Participants) | 1800 | 1331 | 1407 | 1459 | 1208 | 1453 | 3214 | 11872
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Data reported for each substudy/arm separately as some placebo participants were shared among substudies.
  years
    Substudy A: number analyzed (Participants) | 1800 | 0 | 0 | 0 | 0 | 0 | 0 | 1800
    Substudy A | 47 [39 to 56] |  |  |  |  |  |  | 47 [39 to 56]
    Substudy B: number analyzed (Participants) | 0 | 1331 | 0 | 0 | 0 | 0 | 0 | 1331
    Substudy B |  | 47 [38 to 57] |  |  |  |  |  | 47 [38 to 57]
    Substudy C: number analyzed (Participants) | 0 | 0 | 1407 | 0 | 0 | 0 | 0 | 1407
    Substudy C |  |  | 45 [37 to 55] |  |  |  |  | 45 [37 to 55]
    Substudy D: number analyzed (Participants) | 0 | 0 | 0 | 1459 | 0 | 0 | 0 | 1459
    Substudy D |  |  |  | 48 [38 to 58] |  |  |  | 48 [38 to 58]
    Substudy E: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1208 | 0 | 0 | 1208
    Substudy E |  |  |  |  | 50 [40 to 60] |  |  | 50 [40 to 60]
    Substudy F: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1453 | 0 | 1453
    Substudy F |  |  |  |  |  | 52 [41 to 61] |  | 52 [41 to 61]
    Substudy G: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3214 | 3214
    Substudy G |  |  |  |  |  |  | 47 [38 to 57] | 47 [38 to 57]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Data reported for each substudy/arm separately as some placebo participants were shared among substudies.
  Participants
    Substudy A: Sex/Gender: number analyzed (Participants) | 1800 | 0 | 0 | 0 | 0 | 0 | 0 | 1800
    Substudy A: Sex/Gender: Female | 1049 |  |  |  |  |  |  | 1049
    Substudy A: Sex/Gender: Male | 749 |  |  |  |  |  |  | 749
    Substudy A: Sex/Gender: Undifferentiated | 0 |  |  |  |  |  |  | 0
    Substudy A: Sex/Gender: Unknown | 1 |  |  |  |  |  |  | 1
    Substudy A: Sex/Gender: Prefer Not to Answer the Question | 1 |  |  |  |  |  |  | 1
    Substudy B: Sex/Gender: number analyzed (Participants) | 0 | 1331 | 0 | 0 | 0 | 0 | 0 | 1331
    Substudy B: Sex/Gender: Female |  | 755 |  |  |  |  |  | 755
    Substudy B: Sex/Gender: Male |  | 571 |  |  |  |  |  | 571
    Substudy B: Sex/Gender: Undifferentiated |  | 0 |  |  |  |  |  | 0
    Substudy B: Sex/Gender: Unknown |  | 2 |  |  |  |  |  | 2
    Substudy B: Sex/Gender: Prefer Not to Answer the Question |  | 3 |  |  |  |  |  | 3
    Substudy C: Sex/Gender: number analyzed (Participants) | 0 | 0 | 1407 | 0 | 0 | 0 | 0 | 1407
    Substudy C: Sex/Gender: Female |  |  | 875 |  |  |  |  | 875
    Substudy C: Sex/Gender: Male |  |  | 528 |  |  |  |  | 528
    Substudy C: Sex/Gender: Undifferentiated |  |  | 1 |  |  |  |  | 1
    Substudy C: Sex/Gender: Unknown |  |  | 2 |  |  |  |  | 2
    Substudy C: Sex/Gender: Prefer Not to Answer the Question |  |  | 1 |  |  |  |  | 1
    Substudy D: Sex/Gender: number analyzed (Participants) | 0 | 0 | 0 | 1459 | 0 | 0 | 0 | 1459
    Substudy D: Sex/Gender: Female |  |  |  | 871 |  |  |  | 871
    Substudy D: Sex/Gender: Male |  |  |  | 583 |  |  |  | 583
    Substudy D: Sex/Gender: Undifferentiated |  |  |  | 3 |  |  |  | 3
    Substudy D: Sex/Gender: Unknown |  |  |  | 1 |  |  |  | 1
    Substudy D: Sex/Gender: Prefer Not to Answer the Question |  |  |  | 1 |  |  |  | 1
    Substudy E: Sex/Gender: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1208 | 0 | 0 | 1208
    Substudy E: Sex/Gender: Female |  |  |  |  | 794 |  |  | 794
    Substudy E: Sex/Gender: Male |  |  |  |  | 414 |  |  | 414
    Substudy E: Sex/Gender: Undifferentiated |  |  |  |  | 0 |  |  | 0
    Substudy E: Sex/Gender: Unknown |  |  |  |  | 0 |  |  | 0
    Substudy E: Sex/Gender: Prefer Not to Answer the Question |  |  |  |  | 0 |  |  | 0
    Substudy F: Sex/Gender: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1453 | 0 | 1453
    Substudy F: Sex/Gender: Female |  |  |  |  |  | 872 |  | 872
    Substudy F: Sex/Gender: Male |  |  |  |  |  | 581 |  | 581
    Substudy F: Sex/Gender: Undifferentiated |  |  |  |  |  | 0 |  | 0
    Substudy F: Sex/Gender: Unknown |  |  |  |  |  | 0 |  | 0
    Substudy F: Sex/Gender: Prefer Not to Answer the Question |  |  |  |  |  | 0 |  | 0
    Substudy G: Sex/Gender: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3214 | 3214
    Substudy G: Sex/Gender: Female |  |  |  |  |  |  | 2021 | 2021
    Substudy G: Sex/Gender: Male |  |  |  |  |  |  | 1185 | 1185
    Substudy G: Sex/Gender: Undifferentiated |  |  |  |  |  |  | 2 | 2
    Substudy G: Sex/Gender: Unknown |  |  |  |  |  |  | 3 | 3
    Substudy G: Sex/Gender: Prefer Not to Answer the Question |  |  |  |  |  |  | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data reported for each substudy/arm separately as some placebo participants were shared among substudies.
  Participants
    Substudy A: number analyzed (Participants) | 1800 | 0 | 0 | 0 | 0 | 0 | 0 | 1800
    Substudy A: Hispanic or Latino | 186 |  |  |  |  |  |  | 186
    Substudy A: Not Hispanic or Latino | 1614 |  |  |  |  |  |  | 1614
    Substudy A: Unknown or Not Reported | 0 |  |  |  |  |  |  | 0
    Substudy B: number analyzed (Participants) | 0 | 1331 | 0 | 0 | 0 | 0 | 0 | 1331
    Substudy B: Hispanic or Latino |  | 224 |  |  |  |  |  | 224
    Substudy B: Not Hispanic or Latino |  | 1106 |  |  |  |  |  | 1106
    Substudy B: Unknown or Not Reported |  | 1 |  |  |  |  |  | 1
    Substudy C: number analyzed (Participants) | 0 | 0 | 1407 | 0 | 0 | 0 | 0 | 1407
    Substudy C: Hispanic or Latino |  |  | 177 |  |  |  |  | 177
    Substudy C: Not Hispanic or Latino |  |  | 1229 |  |  |  |  | 1229
    Substudy C: Unknown or Not Reported |  |  | 1 |  |  |  |  | 1
    Substudy D: number analyzed (Participants) | 0 | 0 | 0 | 1459 | 0 | 0 | 0 | 1459
    Substudy D: Hispanic or Latino |  |  |  | 311 |  |  |  | 311
    Substudy D: Not Hispanic or Latino |  |  |  | 1147 |  |  |  | 1147
    Substudy D: Unknown or Not Reported |  |  |  | 1 |  |  |  | 1
    Substudy E: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1208 | 0 | 0 | 1208
    Substudy E: Hispanic or Latino |  |  |  |  | 552 |  |  | 552
    Substudy E: Not Hispanic or Latino |  |  |  |  | 656 |  |  | 656
    Substudy E: Unknown or Not Reported |  |  |  |  | 0 |  |  | 0
    Substudy F: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1453 | 0 | 1453
    Substudy F: Hispanic or Latino |  |  |  |  |  | 935 |  | 935
    Substudy F: Not Hispanic or Latino |  |  |  |  |  | 518 |  | 518
    Substudy F: Unknown or Not Reported |  |  |  |  |  | 0 |  | 0
    Substudy G: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3214 | 3214
    Substudy G: Hispanic or Latino |  |  |  |  |  |  | 1467 | 1467
    Substudy G: Not Hispanic or Latino |  |  |  |  |  |  | 1747 | 1747
    Substudy G: Unknown or Not Reported |  |  |  |  |  |  | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data reported for each substudy/arm separately as some placebo participants were shared among substudies.
  Participants
    Substudy A: Race: number analyzed (Participants) | 1800 | 0 | 0 | 0 | 0 | 0 | 0 | 1800
    Substudy A: Race: American Indian or Alaska Native | 19 |  |  |  |  |  |  | 19
    Substudy A: Race: Asian | 35 |  |  |  |  |  |  | 35
    Substudy A: Race: Black, African American, or African | 127 |  |  |  |  |  |  | 127
    Substudy A: Race: Middle Eastern or North African | 81 |  |  |  |  |  |  | 81
    Substudy A: Race: Native Hawaiian or Other Pacific Islander | 3 |  |  |  |  |  |  | 3
    Substudy A: Race: White | 1394 |  |  |  |  |  |  | 1394
    Substudy A: Race: More than one race | 29 |  |  |  |  |  |  | 29
    Substudy A: Race: None of the above | 50 |  |  |  |  |  |  | 50
    Substudy A: Race: Prefer not to answer | 42 |  |  |  |  |  |  | 42
    Substudy A: Race: No response | 20 |  |  |  |  |  |  | 20
    Substudy B: Race: number analyzed (Participants) | 0 | 1331 | 0 | 0 | 0 | 0 | 0 | 1331
    Substudy B: Race: American Indian or Alaska Native |  | 4 |  |  |  |  |  | 4
    Substudy B: Race: Asian |  | 75 |  |  |  |  |  | 75
    Substudy B: Race: Black, African American, or African |  | 96 |  |  |  |  |  | 96
    Substudy B: Race: Middle Eastern or North African |  | 7 |  |  |  |  |  | 7
    Substudy B: Race: Native Hawaiian or Other Pacific Islander |  | 1 |  |  |  |  |  | 1
    Substudy B: Race: White |  | 1041 |  |  |  |  |  | 1041
    Substudy B: Race: More than one race |  | 30 |  |  |  |  |  | 30
    Substudy B: Race: None of the above |  | 43 |  |  |  |  |  | 43
    Substudy B: Race: Prefer not to answer |  | 23 |  |  |  |  |  | 23
    Substudy B: Race: No response |  | 11 |  |  |  |  |  | 11
    Substudy C: Race: number analyzed (Participants) | 0 | 0 | 1407 | 0 | 0 | 0 | 0 | 1407
    Substudy C: Race: American Indian or Alaska Native |  |  | 7 |  |  |  |  | 7
    Substudy C: Race: Asian |  |  | 67 |  |  |  |  | 67
    Substudy C: Race: Black, African American, or African |  |  | 101 |  |  |  |  | 101
    Substudy C: Race: Middle Eastern or North African |  |  | 35 |  |  |  |  | 35
    Substudy C: Race: Native Hawaiian or Other Pacific Islander |  |  | 2 |  |  |  |  | 2
    Substudy C: Race: White |  |  | 1079 |  |  |  |  | 1079
    Substudy C: Race: More than one race |  |  | 23 |  |  |  |  | 23
    Substudy C: Race: None of the above |  |  | 50 |  |  |  |  | 50
    Substudy C: Race: Prefer not to answer |  |  | 33 |  |  |  |  | 33
    Substudy C: Race: No response |  |  | 10 |  |  |  |  | 10
    Substudy D: Race: number analyzed (Participants) | 0 | 0 | 0 | 1459 | 0 | 0 | 0 | 1459
    Substudy D: Race: American Indian or Alaska Native |  |  |  | 10 |  |  |  | 10
    Substudy D: Race: Asian |  |  |  | 92 |  |  |  | 92
    Substudy D: Race: Black, African American, or African |  |  |  | 111 |  |  |  | 111
    Substudy D: Race: Middle Eastern or North African |  |  |  | 59 |  |  |  | 59
    Substudy D: Race: Native Hawaiian or Other Pacific Islander |  |  |  | 5 |  |  |  | 5
    Substudy D: Race: White |  |  |  | 1029 |  |  |  | 1029
    Substudy D: Race: More than one race |  |  |  | 31 |  |  |  | 31
    Substudy D: Race: None of the above |  |  |  | 80 |  |  |  | 80
    Substudy D: Race: Prefer not to answer |  |  |  | 37 |  |  |  | 37
    Substudy D: Race: No response |  |  |  | 5 |  |  |  | 5
    Substudy E: Race: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1208 | 0 | 0 | 1208
    Substudy E: Race: American Indian or Alaska Native |  |  |  |  | 7 |  |  | 7
    Substudy E: Race: Asian |  |  |  |  | 50 |  |  | 50
    Substudy E: Race: Black, African American, or African |  |  |  |  | 104 |  |  | 104
    Substudy E: Race: Middle Eastern or North African |  |  |  |  | 59 |  |  | 59
    Substudy E: Race: Native Hawaiian or Other Pacific Islander |  |  |  |  | 2 |  |  | 2
    Substudy E: Race: White |  |  |  |  | 847 |  |  | 847
    Substudy E: Race: More than one race |  |  |  |  | 31 |  |  | 31
    Substudy E: Race: None of the above |  |  |  |  | 74 |  |  | 74
    Substudy E: Race: Prefer not to answer |  |  |  |  | 27 |  |  | 27
    Substudy E: Race: No response |  |  |  |  | 7 |  |  | 7
    Substudy F: Race: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1453 | 0 | 1453
    Substudy F: Race: American Indian or Alaska Native |  |  |  |  |  | 3 |  | 3
    Substudy F: Race: Asian |  |  |  |  |  | 44 |  | 44
    Substudy F: Race: Black, African American, or African |  |  |  |  |  | 177 |  | 177
    Substudy F: Race: Middle Eastern or North African |  |  |  |  |  | 24 |  | 24
    Substudy F: Race: Native Hawaiian or Other Pacific Islander |  |  |  |  |  | 2 |  | 2
    Substudy F: Race: White |  |  |  |  |  | 1121 |  | 1121
    Substudy F: Race: More than one race |  |  |  |  |  | 17 |  | 17
    Substudy F: Race: None of the above |  |  |  |  |  | 45 |  | 45
    Substudy F: Race: Prefer not to answer |  |  |  |  |  | 16 |  | 16
    Substudy F: Race: No response |  |  |  |  |  | 4 |  | 4
    Substudy G: Race: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3214 | 3214
    Substudy G: Race: American Indian or Alaska Native |  |  |  |  |  |  | 12 | 12
    Substudy G: Race: Asian |  |  |  |  |  |  | 68 | 68
    Substudy G: Race: Black, African American, or African |  |  |  |  |  |  | 433 | 433
    Substudy G: Race: Middle Eastern or North African |  |  |  |  |  |  | 49 | 49
    Substudy G: Race: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  | 4 | 4
    Substudy G: Race: White |  |  |  |  |  |  | 2445 | 2445
    Substudy G: Race: More than one race |  |  |  |  |  |  | 57 | 57
    Substudy G: Race: None of the above |  |  |  |  |  |  | 72 | 72
    Substudy G: Race: Prefer not to answer |  |  |  |  |  |  | 60 | 60
    Substudy G: Race: No response |  |  |  |  |  |  | 14 | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants Randomized Within Each Appendix
Description: Total number of participants randomized within each Appendix will be reported. Appendix-specific outcome measure data will be reported under the associated NCT ID.
Time Frame: Up to approximately 2 years 10 months
Population: Individuals who met inclusion criteria and consented for study drug for each study arm. Given that participants were not randomized at this point, one number is reported for each study arm as a whole.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin
Number analyzed (Participants) | 3457 | 3837 | 3315 | 2212 | 1657 | 1660 | 3704
Participants | 1800 | 1331 | 1407 | 1459 | 1208 | 1453 | 3214

ADVERSE EVENTS:
Time Frame: Up to 180 days
Description: Appendix-specific adverse event data will be reported under the associated NCT ID.
Arm/Group | Arm A - Ivermectin 400 | Arm B - Fluvoxamine | Arm C - Fluticasone | Arm D - Ivermectin 600 | Arm E - Fluvoxamine 100 | Arm F - Montelukast | Arm G - Metformin
All-Cause Mortality (participants affected / at risk) | 0/1800 | 0/1331 | 0/1407 | 0/1459 | 0/1208 | 0/1453 | 0/3214
Serious Adverse Events (participants affected / at risk) | 0/1800 | 0/1331 | 0/1407 | 0/1459 | 0/1208 | 0/1453 | 0/3214
Other Adverse Events (participants affected / at risk) | 0/1800 | 0/1331 | 0/1407 | 0/1459 | 0/1208 | 0/1453 | 0/3214

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT04885530/Prot_SAP_000.pdf